CLINICAL TRIAL: NCT07050667
Title: Treatment of Chronic Wounds With Cold Plasma -Plasma Care® vs. Placebo: a Multicenter, Two-arm, Randomized, Single-blind, Prospective, Clinical Study
Brief Title: Treatment of Chronic Wounds With Cold Plasma -Plasma Care® vs. Placebo
Acronym: SUPCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terraplasma Medical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-2-3/2023; PLASMACARE/70/Q1-23 (Other: LKH Feldkirch)
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hard to Heal Wounds; Infected Wound
Keywords: placebo controlled; plasma care; non thermal plasma; cold atmospheric plasma; wound healing; chronic wounds
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, two-arm, randomized, single-blind, clinical study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma arm (Active Comparator): Treatment of patients with cold atmospheric plasma
  Interventions: Device: Cold atmospheric plasma
- Placebo arm (Placebo Comparator): Placebo control
  Interventions: Device: Placebo treatment

INTERVENTIONS:
Device: Cold atmospheric plasma — Treatment of chronic wounds with cold plasma
  Arms: Plasma arm
Device: Placebo treatment — Treatment of chronic wounds with the placebo device
  Arms: Placebo arm

SUMMARY:
Objective: The study aimed to evaluate the wound healing effects of plasma care®, a cold atmospheric plasma device, in patients with chronic wounds.

Method: A prospective, multicenter, two-arm, randomized, single-blind clinical trial was conducted to compare the effectiveness of plasma care® versus placebo, both combined with best practice wound care.

DETAILED DESCRIPTION:
Chronic wounds present a growing global health challenge, significantly affecting patients' quality of life and imposing high treatment costs. Despite advances in wound care, such as bioactive dressings and specialized medical personnel, effective treatment remains difficult due to the complexity of the wounds and underlying conditions.

Cold atmospheric plasma (CAP) has recently emerged as a promising treatment. CAP is created by ionizing gas with strong electric fields, producing reactive species that stimulate human cell regeneration while also exhibiting strong antibacterial and antifungal effects-even against antibiotic-resistant strains. This dual action makes CAP especially useful for chronic wounds, which are prone to infections.

CAP also benefits wound healing by lowering wound pH. Chronic wounds often have an alkaline environment conducive to bacterial growth, but CAP shifts the pH toward more acidic levels, supporting cell function and antibacterial activity.

Clinical studies have shown CAP significantly improves wound healing by promoting granulation tissue formation, reducing wound size and infection, and alleviating symptoms like redness and itching. CAP has also proven safe, with no mutagenic effects on healthy cells.

Different technologies exist to generate CAP, including Dielectric Barrier Discharge (DBD), Plasma Jet, and Surface Micro Discharge (SMD). The plasma care® device used in this study is based on SMD technology, allowing mobile, gas-free use to treat areas up to 13 cm², with treatment dose determined by application duration.

This study aims to evaluate whether plasma care® provides significantly better healing outcomes in chronic wounds of various types compared to placebo treatment. It also seeks to understand the impact of CAP on wound healing factors such as infection control, pH reduction, and exudate management, alongside patient experiences like pain and tolerability. If successful, this study could establish plasma care® as a valuable new option in chronic wound therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 95 years at the time of consent
* Presence of chronic wounds of any origin and wound phase (Includes locally infected wounds)
* Wound size up to 20 x 10 cm (If multiple wounds are present, one wound is designated as the study wound)

Exclusion Criteria:

* Pregnant and breastfeeding women
* Patients on ongoing systemic antibiotic therapy or who received antibiotics within 1 week prior to study start
* Patients who participated in another study within one month prior to this study
* Patients with acute wounds
* Wounds with visible tendons and bones
* Wounds with more than 30% dry necrosis
* Allergy or intolerance to cold plasma
* Patients with wounds covered by primary or secondary dressings

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Wound area at the end of the study | 42 days
  Size of the wound area (absolute) in cm2
Size and time course of the wound area at the end of the study | 42 days
  Average time course in size (absolute) of the wound area in cm2 per visit
Percentage change in wound area at the end of the study | 42 days
  Wound area as a percentage (from baseline)
Dynamics of the percentage change in wound area from baseline | 42 days
  Average time course of the percentage in wound area (compared to the initial value)

SECONDARY OUTCOMES:
pH value | 42 days
  pH measurement by pH meter
Pain Score | 42 days
  Pain as measured by the VAS Score (1 - 10)
Infection Score | 42 days
  Infection, measured by the PGA - Physician Global Assessment Score ranging from 0 (no signs of infection) to 4 (maximal signs of infection); 1-4 is considered infected
Tolerability of treatment | 42 days
  no problem (e.g. no maceration, deterioration of the wound, blisters) new development/intensification of erythema (maceration, blisters, exudate congestion)
Subjective sensation | 42 days
  Subjective sensation as given by the patient: 1 (pleasant feeling), 2 (no specific sensation), 3 (unpleasant), 4 (very unpleasant)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - LKH Bregenz, Bregenz
  - LKH Feldkirch, Feldkirch

IPD SHARING:
Plan to Share IPD: No
Due to austrian legal privacy laws